CLINICAL TRIAL: NCT03427359
Title: The Efficacy of Induction Chemotherapy With Cisplatin and Capecitabine Followed by Concurrent Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Cisplatin and Capecitabine Followed by Concurrent Chemoradiotherapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O1-HongKongShenzhen
Record Dates: First submitted 2018-01-21; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; induction chemotherapy; cisplatin; capecitabine; chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Capecitabine; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: All patients received 3 cycles of induction chemotherapy (cisplatin 80mg/m2, day 1; oral capecitabine 1000mg/m2 twice daily from day1-14, repeated every 3 weeks) followed by concomitant cisplatin (100mg/m2,day1,every 3 weeks) for a total of 2 cycles with radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Induction chemotherapy: capecitabine tablet 1000mg/m2 po bid from day1 to 14,cisplatin injection 80mg/m2 iv day1,every 3 weeks for a total of 3 cycles. Then followed by concurrent chemoradiotherapy with cisplatin injection 100mg/m2 iv every 3 weeks for a total of 2 cycles.
  Interventions: Drug: cisplatin, capecitabine

INTERVENTIONS:
Drug: cisplatin, capecitabine — Experimental arm patients received 3 cycles of induction chemotherapy (cisplatin 80mg/m2, day 1; oral capecitabine 1000mg/m2 twice daily from day1-14, repeated every 3 weeks) followed by concomitant cisplatin (100mg/m2,day1,every 3 weeks) for a total of 2 cycles with radiotherapy.
  Other Names: chemoradiotherapy

SUMMARY:
To prospectively evaluate the short-term efficacy and toxicity of induction chemotherapy with cisplatin and capecitabine followed by concurrent chemoradiotherapy (CCRT) in the treatment of locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
All patients received 3 cycles of induction chemotherapy:cisplatin 80mg/m2, day 1; oral capecitabine 1000mg/m2 twice daily from day1-14, repeated every 3 weeks followed by concomitant cisplatin (100mg/m2,day1,every 3 weeks) for a total of 2 cycles with radiotherapy. Intensity-modified radiotherapy (IMRT) were used in all patients with the total dose and dose/fraction (Fr) as follows: PTV (planned target volume)_1:70 grays (Gy) at 2 Gy/ Fr, PTV_2:63 Gy at 1.8 Gy/ Fr, PTV_3:56 Gy at 1.6 Gy/ Fr;5 fractions per week. Tumor response was evaluated after 3 cycles of induction chemotherapy and 16 weeks following completion of CCRT according to the Response Evaluation Criteria in Solid Tumors 1.1 (RECIST1.1). All toxicities were gauged based on the Common Terminology Criteria for Adverse Events version 4.03 (CTCAE 4.03).

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed nasopharyngeal carcinoma.
* Staged as III to IVB.
* 18-75 years old.
* Performance status ≤2.
* No previous chemotherapy or radiotherapy.
* No concurrent malignancies or a history of other malignancies.
* Adequate bone marrow function (absolute neutrophil count ≥1.5×109/L, platelets ≥100×109/L).
* Adequate liver and renal function (serum bilirubin and serum transaminase levels less than twice the upper limit of normal, creatinine clearance ≥ 60ml/min).
* Without serious co-morbidity.

Exclusion Criteria:

* Stage I-II or IVC.
* Allergic to cisplatin or capecitabine
* Age <18 or >75
* Performance Status >2.
* Without adequate bone marrow or liver function or renal function.
* Severe co-morbidity and can not tolerate chemotherapy.
* Other conditions not suitable for the study on the discretion of charging doctor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
PFS (progression free survival) | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  progression free survival

IPD SHARING:
Plan to Share IPD: Undecided